# **Official Title:**

Retrospective Evaluation of the Effectiveness of Methotrexate Treatment in Cases with Relative Contraindications in Ectopic Pregnancies

# **NCT Number:**

No

## **Document Date:**

15.05.2025

### INFORMED VOLUNTARY CONSENT FORM

The study you are participating in is a scientific research project titled: "Retrospective Evaluation of the Effectiveness of Methotrexate Treatment in Cases with Relative Contraindications in Ectopic Pregnancies."

#### Aim:

The aim of this study is to reduce the number of patients undergoing surgery due to ectopic pregnancy as much as possible, thereby minimizing the risks associated with anesthesia and surgical complications. By selecting appropriate patients, treatment with methotrexate will both protect the patient from potential complications during anesthesia and surgery and offer a safer and more cost-effective method.

Since this study will be conducted using previously recorded data from the hospital information system, it poses no risk or harm to you. Information such as your age, complaints, obstetric history, blood test results, imaging reports, surgical notes (if applicable), treatment methods, dosage and duration, length of hospital stay, and any blood or blood product transfusions will be collected. This is entirely a statistical and computer-based numerical study and will not harm you. There is no direct benefit or disadvantage to you.

If any development arises during the research that may concern you, this will be immediately communicated to you or your legal representative. If you wish to receive further information about the study or if you experience any issues, side effects, or discomforts related to the study, you can contact **Dr. Gülhan ÖZÜM at 0535....** 

You will not receive any payment for participating in this study; likewise, you will not be charged for any examinations, tests, or medical services related to this study, as only existing test and surgery results will be used.

**Participation in this research is entirely voluntary.** You may refuse to participate or withdraw at any stage without penalty or loss of any benefits. The researcher may also remove you from the study if you fail to comply with its requirements or disrupt the study schedule. The results of this study will be used for scientific purposes; if you withdraw or are removed, your medical data may still be used for scientific purposes if necessary.

All your medical and personal identity information will be kept confidential. Even if the research is published, your identity will not be disclosed. However, authorized research monitors, auditors, ethics committees, and official authorities may access your medical records if required. You may also access your medical information upon request.

### **Consent to Participate in the Study:**

I have read and been verbally informed of the details provided above prior to the commencement of the study. I asked all the questions I had, and I fully understand the explanations given to me both in writing and verbally. I was given sufficient time to decide whether or not I want to participate. Under these conditions, I authorize the researcher to review,

transfer, and process my medical information, and I voluntarily accept the invitation to participate in the study without any pressure or coercion.

A signed copy of this form will be given to me.

| Participant | (Volunteer): |
|-------------------|--------------|
| Name-Surname: | |
| Address: | |
| Phone: | |
| Date & Signature: | |

## **Researcher:**

Name-Surname:

Address:

Phone:

Date & Signature: